CLINICAL TRIAL: NCT06166095
Title: Dose-Response Effect of Exercise on Depression and Brain-Derived Neurotrophic Factor (BDNF) in Sedentary Young Adults
Brief Title: Dose-Response Effect Exercise and Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Central Florida (Other)
Collaborators: American College of Sports Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: STUDY00005112
Record Dates: First submitted 2023-09-28; First posted 2023-12-12 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Depression
Keywords: depression; exercise; BDNF; Brain-derived Neurotrophic Factor; Major Depressive Disorder; MDD
MeSH Terms: conditions — Depression; Motor Activity; Depressive Disorder, Major

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- high-dose moderate to vigorous physical activity (MVPA) (Experimental): Participants will be asked to perform a high-dose (HD) (i.e., 300 minutes of moderate to vigorous physical activity (MVPA) per week) of structured exercise for 10 weeks. Exercise modality and schedule will be participant- selected and may consist of any combination of aerobic and strength training that elevates the heart rate between 64 - 95 percent of estimated heart rate max.
  Participants will be asked to track their activity using Fitbit.
  Interventions: Other: high-dose
- moderate-dose moderate to vigorous physical activity (MVPA) (Experimental): Participants will be asked to perform a moderate-dose (MD) (i.e., 150 minutes of moderate to vigorous physical activity (MVPA) per week) of structured exercise for 10 weeks. Exercise modality and schedule will be participant- selected and may consist of any combination of aerobic and strength training that elevates the heart rate between 64 - 95 percent of estimated heart rate max.
  Participants will be asked to track their activity using Fitbit.
  Interventions: Other: moderate-dose
- walking attention control (Experimental): Participants will be provided sleep education material and will be asked to perform 15 minutes of leisure walking three times per week. This exercise intensity does not meet the recommended volume of exercise necessary for health benefits.
  Instructing participants to walk will reduce the likelihood that participants will undertake a more vigorous exercise routine.
  Participants will be asked to track their sleep each night using Fitbit.
  Interventions: Other: Walking attention control

INTERVENTIONS:
Other: high-dose — Participants will be asked to perform a high-dose (HD) (i.e., 300 minutes of MVPA per week) of structured exercise for 10 weeks. Exercise modality and schedule will be participant- selected and may consist of any combination of aerobic and strength training that elevates the heart rate between 64 - 95 percent of estimated heart rate max
  Arms: high-dose moderate to vigorous physical activity (MVPA)
Other: Walking attention control — The attention control group will be asked to wear the Fitbit activity tracker to monitor their sleep each night for 10 weeks.
  Arms: walking attention control
Other: moderate-dose — Participants will be asked to perform a moderate-dose (MD) (i.e., 150 minutes of MVPA per week) of structured exercise for 10 weeks. Exercise modality and schedule will be participant- selected and may consist of any combination of aerobic and strength training that elevates the heart rate between 64 - 95 percent of estimated heart rate max
  Arms: moderate-dose moderate to vigorous physical activity (MVPA)

SUMMARY:
The present study aims to address gaps in the literature by evaluating the objectively measured dose-response relationship between exercise and depression symptoms; examining changes in resting (Brain-derived Neurotrophic Factor) BDNF from baseline to week 10 of an exercise intervention; and assessing varying exercise intensities on enjoyment, affect, and health-related quality of life in sedentary young adult college students.

DETAILED DESCRIPTION:
This 10-week randomized single-blind controlled trial will consist of an exercise intervention and attention control condition. A two-week familiarity trial period will be followed by 8 weeks of structured exercise. Objectively measured physical activity will be remotely monitored via Fitbit to examine its effect on depressive symptoms in sedentary young adult college students.

Approximately 48 enrolled college students ages 18 - 25 will be recruited for the proposed study and randomized with a 1:1:1 allocation to one of the following conditions:

1. high-dose (HD) moderate to vigorous physical activity (MVPA) (n=16)
2. moderate-dose (MD moderate to vigorous physical activity (MVPA) (n=16)
3. a walking (W) attention control (n=16)

ELIGIBILITY:
Inclusion Criteria:

* enrolled UCF college students aged 18 to 25
* mild to moderate depressive symptoms
* willing to wear a Fitbit for extended periods of time during the study
* willing to participate in moderate-to-vigorous PA
* physically able to participate in exercise safely

Exclusion Criteria:

* under 110 lbs
* history of bad reaction to a past blood draw
* have been advised by a medical provider to not give/donate blood
* presence of anemia
* current cognitive therapy or antidepressant medication
* diagnosis of a co-occurring condition such as attention deficit hyperactivity disorder (ADHD)
* diagnosis of a serious mental illness (SMI) such as schizophrenia or bipolar disorder
* pregnant or nursing
* current smoker
* beta-blocker medications

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2023-07-01 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
Brain-derived Neurotrophic Factor (BDNF) assay | 1 year
  A fasted (> 8 hours) blood draw will be performed at baseline and post-treatment to measure resting serum BDNF levels. Serum concentrations of total BDNF will be measured with Human BDNF Human ELISA assay kits for total serum BDNF from ThermoFisher Scientific

SECONDARY OUTCOMES:
Fitbit for heart rate | 1 year
  Heart rate (bpm.) will be collected through Fitabase from the Fitbit as the participants exercise and/ or walk.
Fitbit for physical activity data | 1 year
  Duration of weekly physical activity (min.) data will be collected from the Fitbit activity trackers.

CONTACTS AND LOCATIONS:
Overall Officials: A'Naja Newsome, PhD, Principal Investigator — University of Central Florida
Locations (1):
- University of Central Florida, Orlando, Florida, United States

IPD SHARING:
Plan to Share IPD: No
Personal information that is collected as part of this research will not be used or distributed for future research studies, even if all identifiers are removed.